CLINICAL TRIAL: NCT04724265
Title: Cytomegalovirus in Perilymphatic Fluid During Cochlear Implantation of Children Presenting a Sensorineural Hearing Loss
Brief Title: Cytomegalovirus (CMV) Perilymphatic Fluid
Acronym: CMVP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191072
Record Dates: First submitted 2021-01-24; First posted 2021-01-26 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Hearing Loss, Cochlear; Cytomegalovirus Congenital
MeSH Terms: conditions — Hearing Loss, Sensorineural; Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collection of sample of perilymphatic fluid during cochlear implantation (Experimental): collection of sample of perilymphatic fluid during cochlear implantation
  Interventions: Biological: collection of sample of perilymphatic fluid during cochlear implantation

INTERVENTIONS:
Biological: collection of sample of perilymphatic fluid during cochlear implantation — collection of sample of perilymphatic fluid during cochlear implantation and to analyse it with a CMV polymerised-chain-reaction to evaluate the involvement of CMV in hearing loss.
  Other Names: collection of perilymphatic fluid

SUMMARY:
In France, children cochlear implantation (CI) is performed 400 times per year. Causes of profound sensorineural hearing loss (SNHL) are represented by congenital malformation of the inner ear for 50 to 60%. Most of the remaining cases of CI in children are caused by congenital CMV infection. The proportion of CMV inducing SNHL with a CI in children is not clearly defined. During CI, we aim to collect a very small sample of perilymphatic fluid and to analyse it with a CMV polymerised-chain-reaction to evaluate the involvement of CMV in SNHL.

DETAILED DESCRIPTION:
Data on etiology of hearing loss and CMV status are collected. Perilymphatic liquid is collected after cochleostomy using a 1ml seringue. The drop of liquid is deposited on a Guthrie card; on another card, a drop of blood is deposited on another card. CMV PCR (polymerised chain reaction) is then performed in order to assess for the presence of CMV. The sensibility, specificity, positive and negative positive values are then calculated.

ELIGIBILITY:
Inclusion Criteria:

* Children (under 18-year-old) presenting with a Sensorineural Hearing Loss with an indication of cochlear implantation

Exclusion Criteria:

-

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of CMV PCR in perilymphatic fluid | 7 days after the collection of the sample (biological collection)
  CMV PCR in perilymphatic fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chebib E, Vauloup-Fellous C, Benoit C, Noel Petroff N, Van Den Abbeele T, Maudoux A, Teissier N. Is CMV PCR of inner ear fluid during cochlear implantation a way to diagnose CMV-related hearing loss? Eur J Pediatr. 2023 Jan;182(1):375-383. doi: 10.1007/s00431-022-04691-6. Epub 2022 Nov 12. PMID 36369401